CLINICAL TRIAL: NCT04250506
Title: A Single-center, Randomized, Double-blind, Placebo- and Moxifloxacin-controlled, Phase 1 Study to Assess the Effect of Single Therapeutic and Supratherapeutic Doses of Daridorexant on the QT Interval Duration in Healthy Subjects
Brief Title: A Study to Assess the Effect of Single Doses of Daridorexant on Electrocardiogram Parameters in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: ID-078-117; 2019-003843-31 (EudraCT Number)
Record Dates: First submitted 2020-01-30; First posted 2020-01-31 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Healthy
MeSH Terms: interventions — daridorexant; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, double-blind, placebo- and moxifloxacin-controlled, Phase 1 study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment A: Daridorexant 50 mg (Experimental): Daridorexant (ACT-541468) administered as film-coated tablets for oral use.
  Interventions: Drug: Daridorexant
- Treatment B: Daridorexant 200 mg (Experimental): Daridorexant (ACT-541468) administered as film-coated tablets (4 x 50 mg) for oral use.
  Interventions: Drug: Daridorexant
- Treatment C: Placebo (Placebo Comparator): Placebo administered as tablets (4 x 50 mg) for oral use.
  Interventions: Drug: Placebo
- Treatment D: Moxifloxacin 400 mg (Active Comparator): Moxifloxacin administered as film-coated tablets for oral use.
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Daridorexant — Daridorexant (ACT-541468) administered as film-coated tablets for oral use.
  Arms: Treatment A: Daridorexant 50 mg; Treatment B: Daridorexant 200 mg
Drug: Placebo — Placebo administered as tablets for oral use.
  Arms: Treatment C: Placebo
Drug: Moxifloxacin — Moxifloxacin administered as film-coated tablets for oral use.
  Arms: Treatment D: Moxifloxacin 400 mg

SUMMARY:
A study to assess the effect of single doses of daridorexant on electrocardiogram parameters in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in the local language prior to any study-mandated procedure.
* Czech citizen with the ability to communicate well with the investigator, in a language understandable to the subject, and to understand and comply with the requirements of the study.
* Healthy male and female subjects aged 18 to 55 years (inclusive) at Screening.
* 12-lead safety ECG: QTcF < 450 ms for male subjects and < 470 ms for female subjects, QRS < 110 ms, and PR < 220 ms, and resting HR > 50 bpm and < 90 bpm with no clinically relevant abnormalities on 12-lead ECG after 5 min in the supine position at Screening and on Day 1 pre-dose of Period 1.
* Healthy on the basis of medical history, physical examination, cardiovascular assessments, and clinical laboratory tests.
* Women of childbearing potential are eligible only if the following applies:

  1. Negative serum pregnancy test at Screening.
  2. Negative serum pregnancy test on Day 1 of the first period.
  3. Agreement to consistently and correctly use a highly effective method of contraception with a failure rate of < 1% per year, be sexually inactive, or have a vasectomized partner from Screening up to at least 30 days after last study treatment administration in the last period with wash-out periods included. If a hormonal contraceptive is used, it must be initiated at least 1 month before first treatment administration.
* Women of non-childbearing potential must meet at least one of the following criteria:

  1. Previous bilateral salpingectomy, salpingo-oophorectomy, or hysterectomy.
  2. Premature ovarian failure confirmed by a specialist gynecologist.
  3. Post-menopausal, defined as 12 consecutive months with amenorrhea prior to Screening without alternative medical cause and confirmed with follicle-stimulating hormone (FSH) test.
  4. XY genotype.
  5. Turner syndrome.
  6. Uterine agenesis.

Exclusion Criteria:

* Pregnant or lactating women.
* Previous exposure to daridorexant.
* Known hypersensitivity to moxifloxacin or any of the drug product excipients or to other fluoroquinolone antibiotics.
* Any contraindication to moxifloxacin treatment.
* History of major medical or surgical disorders which, in the opinion of the investigator, are likely to interfere with the absorption, distribution, metabolism, or excretion of the study treatments (appendectomy and herniotomy allowed, cholecystectomy not allowed).
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* History or presence of rhythm disorders (e.g., sinoatrial heart block, sick-sinus syndrome, second- or third-degree atrioventricular block, long QT syndrome, symptomatic bradycardia, atrial flutter, or atrial fibrillation) or electrolyte disturbances, particularly hypokalemia.
* Any sleep-disorder including self-reported insomnia disorder, breathing-related sleep disorders, restless legs syndrome, nightmare disorder, non-rapid eye movement sleep arousal disorders (sleep terror disorder or sleepwalking disorder), rapid eye movement sleep behavior disorder, circadian rhythm sleep-wake disorders.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-07-22 (Actual)

PRIMARY OUTCOMES:
Placebo-corrected change from baseline in the HR-corrected QTcF (ΔΔQTcF) | Various time points (for up to 24 hours) on Day 1 and Day 2 of each period. The 4 periods will be separated by a wash-out period of 7-10 days. Total duration: up to 8 weeks.

SECONDARY OUTCOMES:
Plasma PK parameters of daridorexant: - AUC from 0 to 24 hours (AUC0-24) | Various time points (for up to 24 hours) on Day 1 and Day 2 of each period. The 4 periods will be separated by a wash-out period of 7-10 days. Total duration: up to 8 weeks.
Plasma PK parameters of daridorexant: - Maximum plasma concentration (Cmax) | Various time points (for up to 24 hours) on Day 1 and Day 2 of each period. The 4 periods will be separated by a wash-out period of 7-10 days. Total duration: up to 8 weeks.
Plasma PK parameters of daridorexant: - Time to reach Cmax (tmax) | Various time points (for up to 24 hours) on Day 1 and Day 2 of each period. The 4 periods will be separated by a wash-out period of 7-10 days. Total duration: up to 8 weeks.
Plasma PK parameters of daridorexant: - T½ | Various time points (for up to 24 hours) on Day 1 and Day 2 of each period. The 4 periods will be separated by a wash-out period of 7-10 days. Total duration: up to 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- CEPHA s.r.o., Pilsen, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schilling U, Henrich A, Muehlan C, Krause A, Dingemanse J, Ufer M. Impact of Daridorexant, a Dual Orexin Receptor Antagonist, on Cardiac Repolarization Following Bedtime Dosing: Results from a Thorough QT Study Using Concentration-QT Analysis. Clin Drug Investig. 2021 Aug;41(8):711-721. doi: 10.1007/s40261-021-01062-1. Epub 2021 Jul 31. PMID 34331678